CLINICAL TRIAL: NCT01586845
Title: A Phase III, Randomized, Multicentre, Open-Label, Concentration-Controlled, Safety and Efficacy Study of Voclosporin and Tacrolimus in Renal Transplantation
Brief Title: Safety and Efficacy Study of Voclosporin and Tacrolimus in Transplantation
Acronym: INSPIRE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ISA10-12
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Renal Transplantation
Keywords: Randomized Controlled Trials; Immunosuppression; Adult; Kidney Transplantation; Treatment Outcome
MeSH Terms: interventions — voclosporin; Tacrolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voclosporin (Experimental): Voclosporin
  Interventions: Drug: voclosporin
- Tacrolimus (Active Comparator): Tacrolimus
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: voclosporin — Initial dose of voclosporin 0.8 mg/kg BID, then concentration controlled
  Other Names: voclosporin, ISA247
  Arms: Voclosporin
Drug: tacrolimus — tacrolimus as per labeled dose
  Arms: Tacrolimus

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of voclosporin administered orally twice daily for the prevention of acute allograft rejection in recipients of a kidney transplant.

DETAILED DESCRIPTION:
This will be a phase III, randomized, multicentre, open-label, concentration-controlled study in subjects undergoing a first or second renal transplant, with induction immunosuppression with an IL-2 receptor antibody (basiliximab), mycophenolate mofetil and steroids.

The primary endpoint to assess non-inferiority will be efficacy failure at the end of Month 12 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-65 years inclusive at the time of screening.
* Recipients of a first or second deceased donor or living donor renal transplant.

Exclusion Criteria:

* Subjects presently receiving immunosuppression for a previously failed transplant.
* Females who are pregnant or nursing or planning to become pregnant during the course of the study, or 3 months after last dose of study medication.
* Sexually-active women of child-bearing potential (including those who are < 1 year postmenopausal) and sexually-active men who are not practicing a highly effective method of birth control.
* Subjects receiving a HLA identical living related transplant.
* Subjects wth a positive T-cell lymphocytotoxic cross match, or positive flow T and B cell cross match.
* Subjects undergoing primary transplant with a current PRA (or CPRA) ≥ 25%.
* Subjects who experienced graft loss within 1 year of transplant.
* Subjects receiving a kidney from a ABO incompatible donor.
* Subjects receiving a kidney from a deceased donor positive for HIV, HBV, HCV or tuberculosis.
* Subjects receiving a a kidney from a non-heart beating donor.
* Subjects receiving paired (en bloc or paired) kidney transplants.
* Transplantation of multiple grafts (e.g. kidney and pancreas).
* Subjects receiving a kidney with a cold ischemia time > 30 hours.
* Subjects receiving any transplanted organ other than a kidney.
* Recipients of a bone marrow or stem cell transplant.
* Any systemic infections requiring continued therapy at the time of entry into this study. (Prophylaxis against CMV and/or PCP infection will be permitted).
* Subjects with positive results of the following serological tests: HIV I Ab, hepatitis B virus (HBV) surface antigen (HBsAg), anti-hepatitis B core antibody (HBcAb), and the anti-hepatitis C virus antibody (HCV Ab). Negative results for these serological tests must be documented within 12 months prior to randomization.
* Subjects with active tuberculosis (Tb) requiring treatment within the last 3 years. Subjects with a known positive purified protein derivative (PPD) test are not eligible unless they have completed treatment for latent Tb and have a negative chest X-ray at time of enrollment. PPD testing must have been done within the last 12 months, and a positive result is defined as ≥ 10 mm induration, a Heaf score of >1 in non-Bacille Calmette-Guérin (BCG) immunized subjects, or >2 in BCG immunized subjects.
* Subjects with a current malignancy or history of malignancy within 5 years or a history of lymphoma at any time. Subjects can be enrolled with a history of squamous or basal cell carcinoma that has been surgically excised or removed with curettage and electrodessication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint to assess non-inferiority will be efficacy failure at the end of Month 12 after randomization. | 1 Year post-Transplant
  FDA Efficacy Failure is biopsy-proven acute rejection (BPAR, Banff Grade ≥ 1A as determined by the central pathologist) where subjects who experience death, graft loss (return to dialysis for >30 days, allograft nephrectomy or re-transplantation), or lost to follow-up are included in the analysis as treatment failures. EMA Efficacy Failure includes any subject experiencing any of the following: biopsy-proven acute rejection (BPAR, Banff Grade ≥ 1A as determined by the central pathologist), death, graft loss or graft dysfunction (Cockcroft-Gault CrCl < 40 mL/min).

REFERENCES:
- [Background] Busque S, Cantarovich M, Mulgaonkar S, Gaston R, Gaber AO, Mayo PR, Ling S, Huizinga RB, Meier-Kriesche HU; PROMISE Investigators. The PROMISE study: a phase 2b multicenter study of voclosporin (ISA247) versus tacrolimus in de novo kidney transplantation. Am J Transplant. 2011 Dec;11(12):2675-84. doi: 10.1111/j.1600-6143.2011.03763.x. Epub 2011 Sep 22. PMID 21943027
- [Background] Kuglstatter A, Mueller F, Kusznir E, Gsell B, Stihle M, Thoma R, Benz J, Aspeslet L, Freitag D, Hennig M. Structural basis for the cyclophilin A binding affinity and immunosuppressive potency of E-ISA247 (voclosporin). Acta Crystallogr D Biol Crystallogr. 2011 Feb;67(Pt 2):119-23. doi: 10.1107/S0907444910051905. Epub 2011 Jan 15. PMID 21245533
- [Background] Birsan T, Dambrin C, Freitag DG, Yatscoff RW, Morris RE. The novel calcineurin inhibitor ISA247: a more potent immunosuppressant than cyclosporine in vitro. Transpl Int. 2005 May;17(12):767-71. doi: 10.1007/s00147-004-0799-z. Epub 2005 Apr 13. PMID 15827754